CLINICAL TRIAL: NCT06975982
Title: Comparison of Symptoms, Pulmonary Function, Muscle Strength, Exercise Capacity, and Frailty Level in Individuals With Esophageal Atresia and Healthy Individuals
Brief Title: Symptoms, Pulmonary Function, Muscle Strength, Exercise Capacity, and Frailty in Esophageal Atresia vs. Healthy Peers
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak-Onal, Principal Investigator, Hacettepe University
Other Study IDs: FTREK24/98
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Atresia; Healthy Children
Keywords: Esophageal atresia; Exercise capacity; Physical activity; Muscle strength
MeSH Terms: conditions — Esophageal Atresia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with esophageal atresia: Children with esophageal atresia
  Interventions: Other: No intervention
- Healthy children: Healthy children
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Esophageal atresia is the most common congenital anomaly of the esophagus and is caused by abnormal development of the esophagus during intrauterine life. In children with esophageal atresia, structural abnormalities due to congenital anomalies and tracheoesophageal fistula, tracheomalacia, respiratory problems, recurrent respiratory tract infections, structural abnormalities, surgical interventions for repair and treatment, and decreased physical activity levels may negatively affect pulmonary function, effective coughing, muscle strength, exercise capacity, posture, motor function, and quality of life. This study aims to compare physical characteristics, body composition, pulmonary function and muscle strength, peak cough flow, posture assessment, peripheral muscle strength test, motor function, exercise capacity, physical activity level, fatigue, frailty and quality of life between children with esophageal atresia and their healthy peers.

ELIGIBILITY:
Esophageal atresia group

Inclusion Criteria:

* Children with esophageal atresia who are willing to participate in the study
* Being between the ages of 6-18,
* Being able to cooperate with the assessments

Exclusion Criteria:

* Being unable to cooperate with the assessments,
* Having an orthopedic, neurological or cardiovascular problem that may affect the assessments,
* Having a lung infection or upper respiratory tract infection in the last four weeks,
* Being an active smoker,
* Not being willing to participate in the study,

Control group

Inclusion Criteria:

* Being between the ages of 6-18,
* Being willing to cooperate with the tests to be performed,
* Being willing to participate in the study.

Exclusion Criteria:

* Having a musculoskeletal problem that may affect exercise performance,
* Having any known chronic disease,
* Having a lung infection or upper respiratory tract infection in the last four weeks,
* Being an active smoker,
* Not willing to participate in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with esophageal atresia and their healthy peers
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-10-24 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Forced expiratory volume in one second | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
Forced expiratory volume in one second/forced vital capacity ratio | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second/forced vital capacity ratio will be recorded.
Peak expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.
Forced mid-expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Forced mid-expiratory flow (FEF25-75) will be recorded.
Body composition | 1st day
  Body composition will be evaluated by triceps skinfold thickness. Skinfold caliper will be used to evaluate triceps skinfold thickness.
Maximal inspiratory pressure | 1st day
  Maximal inspiratory pressure will be measured using an mouthpiece pressure measuring device.
Maximal expiratory pressure | 1st day
  Maximal expiratory pressure will be measured using an mouthpiece pressure measuring device.
Peak cough flow | 1st day
  Peak cough flow will be measured using a peak flow meter.
Hand grip strength | 1st day
  Hand grip strength will be evaluated with a hand dynamometer device.
Knee extensor muscle strength | 1st day
  Knee extensor muscle strength will be assessed with a portable digital dynamometer.
Shoulder abductor muscle strength | 1st day
  Shoulder abductor muscle strength will be assessed with a portable digital dynamometer.
Motor function | 1st day
  Motor function will be assessed using Time Up and Go test. In the Time Up and Go test, the individual is asked to stand up from a standard chair with armrests, walk 3 m, turn, walk back to the chair, and sit down again. The time is recorded in seconds.
Functional exercise capacity | 1st day
  6 minute walk test will be performed to assess functional capacity.
Physical activity level | 1st day
  The Physical Activity Questionnaire for Children (PAQ-C) and the Physical Activity Questionnaire for Adolescents (PAQ-A) will be used to assess physical activity levels. The Turkish versions of these assessment tools have been shown to be valid and reliable. The total score ranges from 1 to 5, where 1 indicates very low physical activity, 5 indicates very high physical activity levels.
Exercise capacity | 1 week after other assessments
  To assess exercise capacity, a symptom-limited cardiopulmonary exercise test will be performed on a bicycle ergometer using Bruce protocol.
Frailty | 1st day
  Frailty level will be calculated using the Composite Frailty Score: (1) Slowness: 6 minute walk test, (2) Weakness: handgrip strength, (3) Fatigue: Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale (PedsQL-MFS), (4) Body composition: triceps skinfold thickness, and (5) Physical activity questionnaire. Each domain is scored on a 0-5 point scale, using z-scores or raw questionnaire scores to assign frailty points (0 = least frail, 5 = most frail). The five domain scores is summed to generate a Composite Frailty Score ranging from 0 to 25, where higher scores reflect greater frailty.

SECONDARY OUTCOMES:
Quality of life assessment | 1st day
  Quality of life will be assessed using Esophageal-Atresia-Quality of Life (EA-QOL) questionnaire. The EA-QOL questionnaire consist of a 17-item parent-reported questionnaire for children aged 2-7 years (eating, physical health and treatment, social isolation, and stress) and a 24-item questionnaire available as child- and parent-reported versions for children aged 8-17 years (eating, social relationships, body image, and health and well-being). Scores range from 0 to 100. Higher scores indicate better quality of life.
Fatigue | 1st day
  Fatigue will be assessed using the Pediatric Quality of Life Multidimensional Fatigue Scale (PedsQL-MFS). The PedsQL-MFS allows the child to assess their own fatigue and parents to assess their child's fatigue. The higher the score, the better the quality of life, indicating fewer fatigue symptoms. Therefore, a score of "0" on the PedsQL-MFS indicates greater fatigue, while a score of "100" indicates less fatigue.
Corbin Posture Rating Scale | 1st day
  Corbin Posture Rating Scale and observational posture analysis. It is an assessment consisting of lateral and posterior posture analysis. '0' is excellent, 12 and above indicates poor posture.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, PhD, PT, Study Director — Hacettepe University; Tutku Soyer, MD, Study Chair — Hacettepe University; Özlem Boybeyi Turer, MD, Study Chair — Hacettepe University; Elmas Ebru Yalcin, MD, Study Chair — Hacettepe University; Nagehan Emiralioglu-Ordukaya, MD, Study Chair — Hacettepe University; Meltem Yildiz-Kayaoglu, MD, Principal Investigator — Hacettepe University; Ismail Songul, MD, Principal Investigator — Hacettepe University; Elif Kocaaga, MSc, PT, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No